CLINICAL TRIAL: NCT02287233
Title: A Phase 1/2 Study of Venetoclax in Combination With Low-Dose Cytarabine in Treatment-Naïve Subjects With Acute Myelogenous Leukemia Who Are ≥ 60 Years of Age and Who Are Not Eligible for Standard Anthracycline-Based Induction Therapy
Brief Title: A Study Evaluating Venetoclax in Combination With Low-Dose Cytarabine in Treatment-Naïve Participants With Acute Myelogenous Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M14-387; 2014-002610-23 (EudraCT Number)
Expanded Access: NCT03123029 (Available)
Record Dates: First submitted 2014-11-06; First posted 2014-11-10 (Estimated); Results first posted 2022-08-29 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Acute Myelogenous Leukemia; AML
Keywords: Myelogenous Leukemia; Treatment Naive AML; Untreated AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myeloid | interventions — venetoclax; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase 1: 600 mg Venetoclax + LDAC (Experimental): Venetoclax was administered orally once daily (QD) on Days 2 through 28 of Cycle 1. Dosing started at 50 mg (Day 2) and increased up to 600 mg by Day 6. Beginning with Cycle 2, 600 mg venetoclax was administered Days 1 through 28 of each 28-day cycle. Participants also received low-dose cytarabine (LDAC; 20 mg/m²) administered by subcutaneous injection once daily on Days 1 to 10 of each cycle.
  Participants could continue receiving treatment until disease progression or until discontinuation criteria were met.
  Interventions: Drug: Venetoclax; Drug: Cytarabine
- Phase 1: 800 mg Venetoclax + LDAC (Experimental): Venetoclax was administered orally once daily (QD) on Days 2 through 28 of Cycle 1. Dosing started at 100 mg (Day 2) and increased up to 800 mg by Day 6. Beginning with Cycle 2, 800 mg venetoclax was administered Days 1 through 28 of each 28-day cycle. Participants also received LDAC (20 mg/m²) administered by subcutaneous injection once daily on Days 1 to 10 of each cycle.
  Participants could continue receiving treatment until disease progression or until discontinuation criteria were met.
  Interventions: Drug: Venetoclax; Drug: Cytarabine
- Phase 2: 600 mg Venetoclax + LDAC (Experimental): Venetoclax was administered orally once daily (QD) on Days 2 through 28 of Cycle 1. Dosing started at 50 mg, and increased up to 600 mg by Day 6. Beginning with Cycle 2, 600 mg venetoclax was administered Days 1 through 28 of each 28-day cycle. Participants also received LDAC (20 mg/m²) administered by subcutaneous injection once daily on Days 1 to 10 of each cycle.
  Participants could continue receiving treatment until disease progression or until discontinuation criteria were met.
  Interventions: Drug: Venetoclax; Drug: Cytarabine

INTERVENTIONS:
Drug: Venetoclax — Venetoclax will be taken orally once daily.
  Other Names: GDC-0199; ABT-199; VENCLEXTA®
Drug: Cytarabine — Low-dose cytarabine will be administered subcutaneously on Days 1 to 10 of each 28-day cycle.

SUMMARY:
This study consists of two parts: A Phase 1 dose-escalation part that will evaluate the safety and pharmacokinetic profile of venetoclax in combination with low-dose cytarabine (LDAC), define the maximum tolerated dose (MTD), and generate data to support a recommended Phase 2 dose (RPTD) in treatment-naïve participants with acute myelogenous leukemia (AML); and a Phase 2 part that will evaluate if the RPTD has sufficient efficacy and acceptable toxicity to warrant further development of the combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be greater than or equal to 65 years of age in Phase 1 and 2. Participants enrolled in Cohort C must be either:

  * greater than or equal to 75 years of age; OR
  * greater than or equal to 60 to 74 years will be eligible if the participants has at least one of the following co-morbidities, which make the participant unfit for intensive chemotherapy:

    * Eastern Cooperative Oncology Group (ECOG) Performance Status of 2 - 3;
    * Cardiac history of congestive heart failure (CHF) requiring treatment or ejection fraction less than or equal to 50% or chronic stable angina;
    * Diffusion capacity of carbon monoxide (DLCO) less than or equal to 65% or forced expiratory volume in one second (FEV1) less than or equal to 65%;
    * Creatinine clearance greater than or equal to 30 mL/min to less than 45 ml/min (calculated by Cockcroft-Gault formula)
    * Moderate hepatic impairment with total bilirubin greater than 1.5 to less than or equal to 3.0 × upper limit of normal (ULN)
    * Any other comorbidity that the physician judges to be incompatible with intensive chemotherapy must be reviewed and approved by the study medical monitor before study enrollment
* Participant must have a projected life expectancy of at least 12 weeks.
* Participant must have histological confirmation of AML and be ineligible for treatment with a standard cytarabine and anthracycline induction regimen due to co-morbidity or other factors.
* Participant must have received no prior treatment for AML with the exception of hydroxyurea, allowed through the first cycle of study treatment. Note: Participant may have been treated for prior Myelodysplastic Syndrome.
* Participant must have an ECOG performance status:

  * of 0 to 2 for participants greater than equal to 75 years of age
  * of 0 to 3 for participants greater than equal to 60 to 74 years of age, if 0 - 1 another co-morbidity is required to make participant eligible.
* Participant must have adequate renal function as demonstrated by a creatinine clearance greater than or equal to 30 mL/min; determined via urine collection for 24-hour creatinine clearance or by the Cockcroft Gault formula.
* Participant must have adequate liver function as demonstrated by:

  * aspartate aminotransferase (AST) less than or equal to 2.5 × ULN
  * alanine aminotransferase (ALT) less than or equal to 2.5 × ULN
  * bilirubin less than or equal to 1.5 × ULN for all participants age 75 and older

    * Participants who are less than 75 years of age must have a bilirubin of less than 3.0 × ULN.

Note: Participants with Gilbert's Syndrome may have a bilirubin greater than 1.5 × ULN per discussion between the investigator and AbbVie medical monitor.

* Male participants must agree to refrain from unprotected sex and sperm donation from initial study drug administration until 180 days after the last dose of study drug.
* Participant must voluntarily sign and date an informed consent, approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to the initiation of any screening or study-specific procedures.
* If female, participant must be either:

  * Postmenopausal defined as no menses for 12 or more months without an alternative medical cause OR
  * Permanently surgical sterile (bilateral oophorectomy, bilateral salpingectomy or hysterectomy)

Exclusion Criteria:

* Participant has received treatment with cytarabine for a pre-existing myeloid disorder.
* Participant has acute promyelocytic leukemia (French-American-British Class M3 AML).
* Participant has known active central nervous system (CNS) involvement with AML.
* Participant has tested positive for human immunodeficiency virus (HIV).
* Participant has received the following within 7 days prior to the initiation of study treatment:

  * Strong and moderate CYP3A inducers such as rifampin, carbamazepine, phenytoin, and St. John's wort.
* Participant has consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges) or Starfruit within 3 days prior to the initiation of study treatment.
* Participant has a cardiovascular disability status of New York Heart Association Class greater than 2.
* Participant has a significant history of renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, hepatic, cardiovascular disease, or any other medical condition that in the opinion of the investigator would adversely affect his/her participating in this study.
* Participant has chronic respiratory disease that requires continuous oxygen use.
* Participant has a malabsorption syndrome or other condition that precludes enteral route of administration.
* Participant exhibits evidence of other clinically significant uncontrolled condition(s) including, but not limited to:

  * Uncontrolled systemic infection requiring intravenous (IV) therapy (viral, bacterial or fungal).
* Participant has a history of other malignancies prior to study entry, with the exception of:

  * Adequately treated in situ carcinoma of the breast or cervix uteri;
  * Basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin;
  * Previous malignancy confined and surgically resected (or treated with other modalities) with curative intent.
* Participant has a white blood cell count greater than 25 × 10^9/L. Note: Hydroxyurea is permitted to meet this criterion.
* Participant is a candidate for a bone marrow or stem cell transplant within 12 weeks after study enrollment.
* Participant has a history of myeloproliferative neoplasm (MPN) including polycythemia vera, myelofibrosis, essential thrombocythemia, or chronic myelogenous leukemia.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2014-12-31 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (9):
- United States (5):
  - Univ Kansas Med Ctr /ID# 131175, Kansas City, Kansas
  - Weill Cornell Medical College /ID# 131170, New York, New York
  - University of Pittsburgh MC /ID# 131168, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center /ID# 131177, Nashville, Tennessee
  - Fred Hutchinson Cancer Research Center /ID# 131178, Seattle, Washington
- Australia (2):
  - Calvary Mater Newcastle /ID# 136076, Waratah, New South Wales
  - Alfred Health /ID# 131180, Melbourne, Victoria
- Universitaetsklinikum Hamburg-Eppendorf (UKE) /ID# 133979, Hamburg, Germany
- Duplicate_A.O.U. Policlinico S.Orsola-Malpighi /ID# 131183, Bologna, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Background] Wei AH, Strickland SA Jr, Hou JZ, Fiedler W, Lin TL, Walter RB, Enjeti A, Tiong IS, Savona M, Lee S, Chyla B, Popovic R, Salem AH, Agarwal S, Xu T, Fakouhi KM, Humerickhouse R, Hong WJ, Hayslip J, Roboz GJ. Venetoclax Combined With Low-Dose Cytarabine for Previously Untreated Patients With Acute Myeloid Leukemia: Results From a Phase Ib/II Study. J Clin Oncol. 2019 May 20;37(15):1277-1284. doi: 10.1200/JCO.18.01600. Epub 2019 Mar 20. PMID 30892988
- [Derived] Wei AH, Panayiotidis P, Montesinos P, Laribi K, Ivanov V, Kim I, Novak J, Champion R, Fiedler W, Pagoni M, Bergeron J, Ting SB, Hou JZ, Yamauchi T, Wang J, Strickland SA, Savona MR, Lin TL, Enjeti AK, Tiong IS, Lee S, Roboz GJ, Popovic R, Jiang Q, Liu Z, Sun Y, Mendes WL, Chyla B, DiNardo CD. Risk stratification of low-dose cytarabine and venetoclax in patients with AML ineligible for intensive chemotherapy. Blood Adv. 2025 Nov 21:bloodadvances.2025017083. doi: 10.1182/bloodadvances.2025017083. Online ahead of print. PMID 41269778
- [Derived] Badawi M, Chen X, Marroum P, Suleiman AA, Mensing S, Koenigsdorfer A, Schiele JT, Palenski T, Samineni D, Hoffman D, Menon R, Salem AH. Bioavailability Evaluation of Venetoclax Lower-Strength Tablets and Oral Powder Formulations to Establish Interchangeability with the 100 mg Tablet. Clin Drug Investig. 2022 Aug;42(8):657-668. doi: 10.1007/s40261-022-01172-4. Epub 2022 Jul 13. PMID 35829925
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — https://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Previously untreated adults with acute myeloid leukemia (AML) who were ineligible for intensive chemotherapy were enrolled at nine study sites in the United States, Australia, Germany, and Italy between December 2014 and May 2017.
  The study consisted of a dose escalation phase (Phase 1) to determine the recommended Phase 2 dose (RPTD), and a dose expansion phase (Phase 2).
Period: Overall Study
Arm/Group | Phase 1: 600 mg Venetoclax + LDAC | Phase 1: 800 mg Venetoclax + LDAC | Phase 2: 600 mg Venetoclax + LDAC
Started | 8 | 10 | 76
Treated | 8 | 10 | 74
Completed (Indicates participants remaining on study) | 0 | 0 | 0
Not Completed | 8 | 10 | 76
Not completed — Adverse Event Not Related to Progression | 1 | 2 | 10
Not completed — Adverse Event Related to Progression | 0 | 2 | 8
Not completed — Physician Decision | 1 | 2 | 4
Not completed — Progressive Disease with Death | 0 | 0 | 10
Not completed — Progressive Disease Without Death | 2 | 3 | 20
Not completed — Withdrawal by Subject | 1 | 1 | 7
Not completed — Other | 3 | 0 | 15
Not completed — Did Not Receive Treatment | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1: 600 mg Venetoclax + LDAC | Phase 1: 800 mg Venetoclax + LDAC | Phase 2: 600 mg Venetoclax + LDAC | Total
Number analyzed (Participants) | 8 | 10 | 76 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.3 (6.45) | 74.4 (3.72) | 75.0 (5.56) | 74.9 (5.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 27 | 33
  Male | 5 | 7 | 49 | 61
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 8 | 10 | 69 | 87
  Black or African American | 0 | 0 | 2 | 2
  Asian | 0 | 0 | 2 | 2
  Missing | 0 | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants With Dose-limiting Toxicities
Description: Dose-limiting toxicities (DLTs) were determined during cycle 1 of the dose-escalation phase and defined as Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 grade 4 (life threatening requiring urgent intervention) or 5 (resulted in death) toxicity, excluding adverse events commonly caused by AML (eg, neutropenia, fever). Hematologic DLT was defined as failure of platelet recovery to 25 × 10^9/L or greater and absolute neutrophil count (ANC) to 0.5 × 10^9/L or greater within 14 days of the last dose of venetoclax in the absence of residual AML.
Time Frame: Up to 28 days (Cycle 1)
Population: The DLT-evaluable population included participants who received at least 80% of planned Cycle 1 doses during the dose-escalation phase (Phase 1)
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1: 600 mg Venetoclax + LDAC: Venetoclax was administered orally once daily (QD) on Days 2 through 28 of Cycle 1. Dosing started at 50 mg (Day 2) and increased up to 600 mg by Day 6. Beginning with Cycle 2, 600 mg venetoclax was administered Days 1 through 28 of each 28-day cycle. Participants also received low-dose cytarabine (LDAC; 20 mg/m²) administered by subcutaneous injection once daily on Days 1 to 10 of each cycle.
- Phase 1: 800 mg Venetoclax + LDAC: Venetoclax was administered orally once daily (QD) on Days 2 through 28 of Cycle 1. Dosing started at 100 mg (Day 2) and increased up to 800 mg by Day 6. Beginning with Cycle 2, 800 mg venetoclax was administered Days 1 through 28 of each 28-day cycle. Participants also received LDAC (20 mg/m²) administered by subcutaneous injection once daily on Days 1 to 10 of each cycle.
Arm/Group | Phase 1: 600 mg Venetoclax + LDAC | Phase 1: 800 mg Venetoclax + LDAC
Number analyzed (Participants) | 8 | 10
Participants | 0 | 1

2. Primary Outcome: Phase 1: Maximum Observed Plasma Concentration (Cmax) of Venetoclax
Description: The highest concentration that a drug achieves in the blood after administration in a dosing interval.
Time Frame: Cycle 1, Day 10 at predose and 2, 4, 6, 8, and 24 hours postdose (venetoclax with LDAC); Cycle 1, Day 18 at predose, 2, 4, 6, 8, and 24 hours postdose (venetoclax alone)
Population: Participants enrolled in Phase 1 who had at least one dose of venetoclax and had at least one reported pharmacokinetic (PK) sample concentration.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Phase 1: 600 mg Venetoclax + LDAC | Phase 1: 800 mg Venetoclax + LDAC
Number analyzed (Participants) | 7 | 10
µg/mL
  Cycle 1, Day 10 (Venetoclax with LDAC) | 2.04 (1.45) | 2.26 (0.930)
  Cycle 1, Day 18 (Venetoclax alone) | 2.92 (2.15) | 2.36 (1.22)

3. Primary Outcome: Phase 1: Time to Maximum Observed Plasma Concentration (Tmax) of Venetoclax
Description: The time at which the maximum plasma concentration (Cmax) is observed.
Time Frame: as for outcome 2
Population: Participants enrolled in Phase 1 who had at least one dose of venetoclax and had at least one reported PK sample concentration
Measure: Median (Full Range); unit: hours
Arm/Group | Phase 1: 600 mg Venetoclax + LDAC | Phase 1: 800 mg Venetoclax + LDAC
Number analyzed (Participants) | 7 | 10
hours
  Cycle 1, Day 10 (Venetoclax with LDAC) | 4.0 [4.0 to 6.0] | 8.0 [4.0 to 8.0]
  Cycle 1, Day 18 (Venetoclax Alone) | 7.0 [3.5 to 8.0] | 6.6 [4.0 to 8.0]

4. Primary Outcome: Phase 1: Area Under the Plasma Concentration-Time Curve Over Time From 0 to 24 Hours (AUC0-24) of Venetoclax
Time Frame: as for outcome 2
Population: Participants enrolled in Phase 1 who had at least one dose of venetoclax and had at least one reported PK sample concentration with available data at each time point
Measure: Mean (Standard Deviation); unit: µg*h/mL
Arm/Group | Phase 1: 600 mg Venetoclax + LDAC | Phase 1: 800 mg Venetoclax + LDAC
Number analyzed (Participants) | 7 | 10
µg*h/mL
  Cycle 1, Day 10 (Venetoclax with LDAC) | 33.3 (27.5) | 33.4 (14.1)
  Cycle 1, Day 18 (Venetoclax Alone): number analyzed (Participants) | 6 | 9
  Cycle 1, Day 18 (Venetoclax Alone) | 51.8 (36.9) | 35.4 (19.8)

5. Primary Outcome: Phase 1: Maximum Observed Plasma Concentration (Cmax) of Cytarabine
Description: The highest concentration that a drug achieves in the blood after administration in a dosing interval.
Time Frame: Cycle 1, Day 1 and Day 10 at pre-dose and at 15 and 30 minutes and 1, 3, 6 hours post-dose.
Population: Participants enrolled in Phase 1 who had at least one dose of cytarabine and had at least one reported PK sample concentration.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 1: 600 mg Venetoclax + LDAC | Phase 1: 800 mg Venetoclax + LDAC
Number analyzed (Participants) | 7 | 10
ng/mL
  Cycle 1, Day 1 (LDAC Alone) | 175 (47.0) | 174 (55.4)
  Cycle 1, Day 10 (LDAC with Venetoclax) | 166 (32.1) | 175 (62.3)

6. Primary Outcome: Phase 1: Time to Maximum Observed Plasma Concentration (Tmax) of Cytarabine
Description: The time at which the maximum plasma concentration (Cmax) is observed.
Time Frame: Cycle 1, Day 1 and Day 10 at pre-dose and at 15 and 30 minutes and 1, 3, 6 hours post-dose.
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | Phase 1: 600 mg Venetoclax + LDAC | Phase 1: 800 mg Venetoclax + LDAC
Number analyzed (Participants) | 7 | 10
hours
  Cycle 1, Day 1 (LDAC Alone) | 0.3 [0.3 to 0.4] | 0.3 [0.2 to 0.5]
  Cycle 1, Day 10 (LDAC with Venetoclax) | 0.3 [0.3 to 0.5] | 0.3 [0.2 to 0.5]

7. Primary Outcome: Phase 1: Area Under the Plasma Concentration-Time Curve Over Time From 0 to Last Measurable Concentration (AUCt) of Cytarabine
Time Frame: Cycle 1, Day 1 and Day 10 at pre-dose and at 15 and 30 minutes and 1, 3, 6 hours post-dose.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Phase 1: 600 mg Venetoclax + LDAC | Phase 1: 800 mg Venetoclax + LDAC
Number analyzed (Participants) | 7 | 10
ng*h/mL
  Cycle 1, Day 1 (LDAC Alone) | 194 (66.3) | 204 (62.9)
  Cycle 1, Day 10 (LDAC with Venetoclax) | 231 (89.0) | 202 (54.9)

8. Primary Outcome: Overall Response Rate
Description: Overall response rate (ORR) is defined as the percentage of participants who achieved a complete remission (CR), complete remission with incomplete marrow recovery (CRi), or partial remission (PR) per the International Working Group (IWG) for AML response criteria, per investigator assessment.
  CR: absolute neutrophil count (ANC) ≥ 10^3 /µL, platelet counts ≥ 10^5 /µL, red blood cell (RBC) transfusion independence (a period of at least 56 days with no RBC transfusion), and bone marrow with < 5% blasts.
  CRi: lack of morphologic evidence of leukemia (blasts < 5%), and platelet counts < 10^5 /µL or ANC < 10^3 /µL.
  PR: all of the hematologic values for a CR but with a decrease of at least 50% in the percentage of blasts to 5% to 25% in the bone marrow aspirate.
Time Frame: Response was assessed at Cycle 2, Day 1, Cycle 4, Day 1, and every 3 cycles thereafter; median duration of treatment was 4.2 months.
Population: All enrolled participants who received venetoclax with LDAC at the recommended Phase 2 dose (600 mg). Efficacy endpoints were pre-specified for Phase 2 only, and are reported for all participants who received the RPTD.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase 1+2: 600 mg Venetoclax + LDAC: Venetoclax was administered orally once daily (QD) on Days 2 through 28 of Cycle 1. Dosing started at 50 mg, and increased up to 600 mg by Day 6. Beginning with Cycle 2, 600 mg venetoclax was administered Days 1 through 28 of each 28-day cycle. Participants also received LDAC (20 mg/m²) administered by subcutaneous injection once daily on Days 1 to 10 of each cycle.
  Participants could continue receiving treatment until disease progression or until discontinuation criteria were met.
Arm/Group | Phase 1+2: 600 mg Venetoclax + LDAC
Number analyzed (Participants) | 82
percentage of participants | 54.9 [43.5 to 65.9]

9. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. The investigator rated the severity of each AE according to the CTCAE Version 4.0 and the following:
  Grade 1: The AE is transient and easily tolerated (mild).
  Grade 2: The AE causes discomfort and interrupts usual activities (moderate).
  Grade 3: The AE causes considerable interference with usual activities and may be incapacitating (moderate to severe).
  Grade 4: The AE is life threatening requiring urgent intervention.
  Grade 5: The AE resulted in death.
  The investigator assessed each event as either having a reasonable possibility or no reasonable possibility of being related to the use of study drug.
  Treatment-emergent events are defined as events that began or worsened in severity after the first dose of study drug.
Time Frame: From first dose of study drug until 30 days after last dose of study drug; median (minimum, maximum) duration of treatment was 4.1 (0.2, 62.8) months overall.
Population: All enrolled participants who received at least one dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: 600 mg Venetoclax + LDAC | Phase 1: 800 mg Venetoclax + LDAC | Phase 2: 600 mg Venetoclax + LDAC
Number analyzed (Participants) | 8 | 10 | 74
Participants
  Any treatment-emergent adverse event (TEAE) | 8 | 10 | 74
  TEAE with CTCAE Grade 3 or 4 | 8 | 10 | 72
  TEAE with CTCAE Grade 3 or above | 8 | 10 | 72
  Venetoclax-related TEAE | 8 | 9 | 66
  LDAC-related TEAE | 8 | 9 | 71
  TEAE leading to hospitalization | 7 | 8 | 64
  TEAE leading to venetoclax discontinuation | 3 | 5 | 24
  TEAE leading to LDAC discontinuation | 3 | 5 | 26
  TEAE leading to venetoclax interruption | 3 | 4 | 45
  TEAE leading to LDAC interruption | 3 | 3 | 38
  TEAE leading to venetoclax reduction | 0 | 1 | 6
  TEAE leading to LDAC reduction | 0 | 0 | 1
  TEAE leading to death | 1 | 4 | 15

10. Secondary Outcome: Complete Remission Rate
Description: Complete remission (CR) rate is defined as the percentage of participants who achieved a complete remission at any time point during the study per the modified IWG criteria for AML and investigator assessment.
  CR: absolute neutrophil count (ANC) ≥ 10^3 /µL, platelet counts ≥ 10^5 /µL, red blood cell (RBC) transfusion independence (a period of at least 56 days with no RBC transfusion), and bone marrow with < 5% blasts.
  Participants who never achieved CR or had no IWG disease assessment were considered to be non-responders in the calculation of CR rate.
Time Frame: as for outcome 8
Population: All enrolled participants who received venetoclax with LDAC at the recommended Phase 2 dose (600 mg)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1+2: 600 mg Venetoclax + LDAC
Number analyzed (Participants) | 82
percentage of participants | 25.6 [16.6 to 36.4]

11. Secondary Outcome: Complete Remission Plus CR With Incomplete Blood Count Recovery (CRi) Rate
Description: The percentage of participants who achieved a CR or CRi at any time point during the study per the modified IWG criteria for AML and investigator assessment.
  CR: absolute neutrophil count (ANC) ≥ 10^3 /µL, platelet counts ≥ 10^5 /µL, red blood cell (RBC) transfusion independence (a period of at least 56 days with no RBC transfusion), and bone marrow with < 5% blasts.
  CRi: lack of morphologic evidence of leukemia (blasts < 5%), and platelet counts < 10^5 /µL or ANC < 10^3 /µL
  Participants who never achieved CR or CRi or had no IWG disease assessment were considered to be non-responders in the calculation of CR + CRi rate.
Time Frame: as for outcome 8
Population: All enrolled participants who received venetoclax with LDAC at the recommended Phase 2 dose (600 mg)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1+2: 600 mg Venetoclax + LDAC
Number analyzed (Participants) | 82
percentage of participants | 53.7 [42.3 to 64.7]

12. Secondary Outcome: CR Plus CRi Rate by Initiation of Cycle 2
Description: The percentage of participants who achieved a CR or CRi by initiation of Cycle 2 of study treatment per the modified IWG criteria for AML and investigator assessment.
  CR: ANC ≥ 10^3 /µL, platelet counts ≥ 10^5 /µL, RBC transfusion independence (a period of at least 56 days with no RBC transfusion), and bone marrow with < 5% blasts.
  CRi: Lack of morphologic evidence of leukemia (blasts < 5%), and platelet counts < 10^5 /µL or ANC < 10^3 /µL.
  Participants who never achieved CR or CRi or had no IWG disease assessment by initiation of Cycle 2 were considered to be non-responders in the calculation of CR + CRi rate by initiation of Cycle 2.
Time Frame: Cycle 2, Day 1
Population: All enrolled participants who received venetoclax with LDAC at the recommended Phase 2 dose (600 mg)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1+2: 600 mg Venetoclax + LDAC
Number analyzed (Participants) | 82
percentage of participants | 28.0 [18.7 to 39.1]

13. Secondary Outcome: Time to First Response of CR + CRi
Description: The time to the first response of CR + CRi is defined as the time from the first date of study drug to the first response of CR or CRi per the IWG AML response criteria assessed by the investigator.
  CR: absolute neutrophil count (ANC) ≥ 10^3 /µL, platelet counts ≥ 10^5 /µL, RBC transfusion independence (a period of at least 56 days with no RBC transfusion), and bone marrow with < 5% blasts.
  CRi: lack of morphologic evidence of leukemia (blasts < 5%), and platelet counts < 10^5 /µL or ANC < 10^3 /µL.
Time Frame: as for outcome 8
Population: Enrolled participants who received venetoclax with LDAC at the recommended Phase 2 dose (600 mg) with a response of CR or CRi
Measure: Median (Full Range); unit: months
Arm/Group | Phase 1+2: 600 mg Venetoclax + LDAC
Number analyzed (Participants) | 44
months | 1.4 [0.8 to 14.9]

14. Secondary Outcome: Time to Best Response of CR + CRi
Description: The time to the best response of CR + CRi is defined as the time from the first date of study drug to the best response of CR or CRi per the IWG AML response criteria assessed by the investigator.
  CR: absolute neutrophil count (ANC) ≥ 10^3 /µL, platelet counts ≥ 10^5 /µL, RBC transfusion independence (a period of at least 56 days with no RBC transfusion), and bone marrow with < 5% blasts.
  CRi: lack of morphologic evidence of leukemia (blasts < 5%), and platelet counts < 10^5 /µL or ANC < 10^3 /µL.
Time Frame: as for outcome 8
Population: as for outcome 13
Measure: Median (Full Range); unit: months
Arm/Group | Phase 1+2: 600 mg Venetoclax + LDAC
Number analyzed (Participants) | 44
months | 2.8 [0.8 to 22.4]

15. Secondary Outcome: Complete Remission With Partial Hematologic Recovery (CRh) Rate
Description: Complete remission with partial hematologic recovery is a derived response based on bone marrow blast and hematology laboratory values. CRh rate is defined as the percentage of participants who achieved CRh as the best response at any time point during the study.
  A participant achieved a CRh when meeting the following criteria:
  * Bone marrow with < 5% blasts and
  * Peripheral blood neutrophil count of > 0.5 × 10^3 /µL and
  * Peripheral blood platelet count of > 0.5 × 10^5 /µL and
  * A 1 week (≥ 7 days) platelet transfusion-free period prior to the hematology lab collection.
  Participants who never achieved CRh or did not have disease assessment or hematology data were considered to be non-responders in the calculation of CRh rate.
Time Frame: as for outcome 8
Population: All enrolled participants who received venetoclax with LDAC at the recommended Phase 2 dose (600 mg)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1+2: 600 mg Venetoclax + LDAC
Number analyzed (Participants) | 82
percentage of participants | 20.7 [12.6 to 31.1]

16. Secondary Outcome: CR Plus CRh Rate
Description: CR + CRh rate is defined as the percentage of participants who achieved CR or CRh at any time point during the study.
  CR: ANC ≥ 10^3 /µL, platelet counts ≥ 10^5 /µL, RBC transfusion independence (a period of at least 56 days with no RBC transfusion), and bone marrow with < 5% blasts.
  CRh is a derived response based on bone marrow blast and hematology lab values. A participant achieved a CRh when meeting the following criteria:
  * Bone marrow with < 5% blasts and
  * Peripheral blood neutrophil count of > 0.5 × 10^3 /µL and
  * Peripheral blood platelet count of > 0.5 × 10^5 /µL and
  * A 1 week (≥ 7 days) platelet transfusion-free period prior to the hematology lab collection.
  Participants who never achieved CR/CRh or did not have disease assessment or hematology data were considered to be non-responders in the calculation of CR + CRh rate.
Time Frame: as for outcome 8
Population: All enrolled participants who received venetoclax with LDAC at the recommended Phase 2 dose (600 mg)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1+2: 600 mg Venetoclax + LDAC
Number analyzed (Participants) | 82
percentage of participants | 46.3 [35.3 to 57.7]

17. Secondary Outcome: CR Plus CRh Rate by Initiation of Cycle 2
Description: CR + CRh rate by initiation of Cycle 2 is defined as the percentage of participants who achieved CR or CRh by initiation of Cycle 2 of study treatment.
  CR: ANC ≥ 10^3 /µL, platelet counts ≥ 10^5 /µL, RBC transfusion independence (a period of at least 56 days with no RBC transfusion), and bone marrow with < 5% blasts.
  CRh is a derived response based on bone marrow blast and hematology lab values. A participant achieved a CRh when meeting the following criteria:
  * Bone marrow with < 5% blasts and
  * Peripheral blood neutrophil count of > 0.5 × 10^3 /µL and
  * Peripheral blood platelet count of > 0.5 × 10^5 /µL and
  * A 1 week (≥ 7 days) platelet transfusion-free period prior to the hematology lab collection.
  Participants who never achieved CR/CRh or did not have disease assessment by initiation of Cycle 2 were considered to be non-responders in the calculation of CR + CRh rate by initiation of Cycle 2.
Time Frame: Cycle 2, Day 1
Population: All enrolled participants who received venetoclax with LDAC at the recommended Phase 2 dose (600 mg)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1+2: 600 mg Venetoclax + LDAC
Number analyzed (Participants) | 82
percentage of participants | 30.5 [20.8 to 41.6]

18. Secondary Outcome: Time to First Response of CR Plus CRh
Description: The time to the first response of CR + CRh is defined as the time from the first date of study drug to the first response of CR or CRh.
  CR: ANC ≥ 10^3 /µL, platelet counts ≥ 10^5 /µL, RBC transfusion independence (a period of at least 56 days with no RBC transfusion), and bone marrow with < 5% blasts.
  CRh is a derived response based on bone marrow blast and hematology lab values. A participant achieved a CRh when meeting the following criteria:
  * Bone marrow with < 5% blasts and
  * Peripheral blood neutrophil count of > 0.5 × 10^3 /µL and
  * Peripheral blood platelet count of > 0.5 × 10^5 /µL and
  * A 1 week (≥ 7 days) platelet transfusion-free period prior to the hematology lab collection.
Time Frame: as for outcome 8
Population: Enrolled participants who received venetoclax with LDAC at the recommended Phase 2 dose (600 mg) with a response of CR or CRh
Measure: Median (Full Range); unit: months
Arm/Group | Phase 1+2: 600 mg Venetoclax + LDAC
Number analyzed (Participants) | 38
months | 1.0 [0.8 to 9.4]

19. Secondary Outcome: Time to Best Response of CR Plus CRh
Description: The time to the best response of CR + CRh is defined as the time from the first date of study drug to the best response of CR or CRh.
  CR: ANC ≥ 10^3 /µL, platelet counts ≥ 10^5 /µL, RBC transfusion independence (a period of at least 56 days with no RBC transfusion), and bone marrow with < 5% blasts.
  CRh is a derived response based on bone marrow blast and hematology lab values. A participant achieved a CRh when meeting the following criteria:
  * Bone marrow with < 5% blasts and
  * Peripheral blood neutrophil count of > 0.5 × 10^3 /µL and
  * Peripheral blood platelet count of > 0.5 × 10^5 /µL and
  * A 1 week (≥ 7 days) platelet transfusion-free period prior to the hematology lab collection.
Time Frame: as for outcome 8
Population: as for outcome 18
Measure: Median (Full Range); unit: months
Arm/Group | Phase 1+2: 600 mg Venetoclax + LDAC
Number analyzed (Participants) | 38
months | 2.6 [0.8 to 22.4]

20. Secondary Outcome: Best Response Based on IWG Criteria
Description: Best response determined using the IWG-AML response criteria during the course of treatment.
  * CR: ANC ≥ 10^3 /µL, platelet counts ≥ 10^5 /µL, RBC transfusion independence, and bone marrow with < 5% blasts;
  * CRi: lack of morphologic evidence of leukemia (blasts < 5%), and platelet counts < 10^5 /µL or ANC < 10^3 /µL;
  * PR: all of the hematologic values for a CR but with a decrease of at least 50% in the percentage of blasts to 5% to 25% in the bone marrow aspirate;
  * MLFS: < 5% blasts in an aspirate and/or bone marrow core sample;
  * RD: failure to achieve CR, CRi, PR; only including subjects surviving at least 7 days following completion of initial treatment cycle with evidence of persistent leukemia by blood and/or bone marrow examination;
  * PD: one or more of the following: ≥ 50% decrement from maximum response levels in neutrophils or platelets; a reduction in hemoglobin by at least 2 g/dL; or transfusion dependence not due to other toxicities and bone marrow blast ≥ 5%.
Time Frame: as for outcome 8
Population: All enrolled participants who received venetoclax with LDAC at the recommended Phase 2 dose (600 mg)
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1+2: 600 mg Venetoclax + LDAC
Number analyzed (Participants) | 82
Participants
  Complete Remission (CR) | 21
  Complete Remission with Incomplete Marrow Recovery (CRi) | 23
  Partial Remission (PR) | 1
  Morphologically Leukemia Free State (MLFS) | 6
  Resistant Disease (RD) | 19
  Disease Progression (PD) | 4
  Discontinued With No Response Data (DS) | 8

21. Secondary Outcome: Duration of Complete Response
Description: Duration of CR is defined as the time from date that a participant achieved CR to the first date of relapse, clinical disease progression or death due to disease progression, whichever occurred earliest. Duration of CR was estimated using Kaplan-Meier methodology. If a participant was still responding at the data cutoff date, then the participant's data were censored at their last disease assessment date. Disease assessment data after the onset of any post-treatment therapy were not included in the duration of CR analysis.
Time Frame: Median duration of follow-up was 44.5 months (range: 0.3 to 63.7)
Population: Enrolled participants who received venetoclax with LDAC at the recommended Phase 2 dose (600 mg) with a response of CR
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1+2: 600 mg Venetoclax + LDAC
Number analyzed (Participants) | 21
months | 14.8 [7.2 to NA] — Could not be estimated due to the low number of events

22. Secondary Outcome: Duration of CR Plus CRi
Description: Duration of CR + CRi is defined as the time from the date that a participant achieved CR or CRi to the first date of relapse, clinical disease progression or death due to disease progression, whichever occurred earliest. Duration of CR + CRi was estimated using Kaplan-Meier methodology. If a participant was still responding at the data cutoff date, then the participant's data were censored at their last disease assessment date. Disease assessment data after the onset of any post-treatment therapy were not included in the analysis.
Time Frame: Median duration of follow-up was 44.5 months (range: 0.3 to 63.7)
Population: as for outcome 13
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1+2: 600 mg Venetoclax + LDAC
Number analyzed (Participants) | 44
months | 9.8 [5.3 to 14.9]

23. Secondary Outcome: Duration of CRi
Description: Duration of CRi is defined as the time from date that a participant achieved CRi to the first date of relapse, clinical disease progression or death due to disease progression, whichever occurred earliest. Duration of CRi was estimated using Kaplan-Meier methodology. If a participant was still responding at the data cutoff date, then the participant's data were censored at their last disease assessment date. Disease assessment data after the onset of any post-treatment therapy were not included in the analysis.
Time Frame: Median duration of follow-up was 44.5 months (range: 0.3 to 63.7)
Population: Enrolled participants who received venetoclax with LDAC at the recommended Phase 2 dose (600 mg) with a response of CRi
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1+2: 600 mg Venetoclax + LDAC
Number analyzed (Participants) | 23
months | 4.7 [2.6 to 5.6]

24. Secondary Outcome: Duration of CR Plus CRh
Description: Duration of CR + CRh is defined as the time from date that a participant achieved CR or CRh to the first date of relapse, clinical disease progression or death due to disease progression, whichever occurred earliest. Duration of CR + CRh was estimated using Kaplan-Meier methodology. If a participant was still responding at the data cutoff date, then the participant's data were censored at their last disease assessment date. Disease assessment data after the onset of any post-treatment therapy were not included in the analysis.
Time Frame: Median duration of follow-up was 44.5 months (range: 0.3 to 63.7)
Population: as for outcome 18
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1+2: 600 mg Venetoclax + LDAC
Number analyzed (Participants) | 38
months | 11.0 [6.1 to 28.2]

25. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from the date of first dose to the date of death. All events of death were included, regardless of whether the event occurred while the participant was still taking study drug, or after the participant discontinued study drug. OS was estimated using Kaplan-Meier methodology. Participants who were still alive were censored at the analysis date.
Time Frame: Median duration of follow-up was 44.5 months (range: 0.3 to 63.7)
Population: Enrolled participants who received venetoclax with LDAC at the recommended Phase 2 dose (600 mg)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1+2: 600 mg Venetoclax + LDAC
Number analyzed (Participants) | 82
months | 9.7 [5.7 to 14.0]

26. Secondary Outcome: Post Baseline Transfusion Independence Rate
Description: Post baseline transfusion independence rate was estimated as the percentage of participants who achieved transfusion independence during the evaluation period. Post-baseline transfusion independence is defined as a period of at least 56 days (≥ 56 days) with no RBC or platelet transfusion during the evaluation period. The evaluation period is from the first dose of study drug to the last dose of study drug until the 30 day follow-up visit, disease progression (including clinical progression), or death, whichever was earlier.
  Results are reported for participants who achieved both RBC and platelet transfusion independence and for participants who received RBC transfusion independence and platelet transfusion independence.
Time Frame: From the first dose of study drug to the last dose of study drug plus 30 days, disease progression (including clinical progression), or death, whichever was earlier; median duration of treatment was 4.2 months.
Population: Enrolled participants who received venetoclax with LDAC at the recommended Phase 2 dose (600 mg)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1+2: 600 mg Venetoclax + LDAC
Number analyzed (Participants) | 82
percentage of participants
  RBC and platelet transfusion independence | 45.1 [34.1 to 56.5]
  RBC transfusion independence | 47.6 [36.4 to 58.9]
  Platelet transfusion independence | 58.5 [47.1 to 69.3]

27. Secondary Outcome: Post Baseline Transfusion Independence Rate Among Participants Transfusion-dependent at Baseline
Description: as for outcome 26
Time Frame: as for outcome 26
Population: Enrolled participants who received venetoclax with LDAC at the recommended Phase 2 dose (600 mg) who received a RBC or platelet transfusion within 8 weeks prior to first dose (60), an RBC transfusion within 8 weeks prior to first dose (53) or a platelet transfusion within 8 weeks prior to first dose (23).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1+2: 600 mg Venetoclax + LDAC
Number analyzed (Participants) | 60
percentage of participants
  RBC and platelet transfusion independence | 45.0 [32.1 to 58.4]
  RBC transfusion independence: number analyzed (Participants) | 53
  RBC transfusion independence | 45.3 [31.6 to 59.6]
  Platelet transfusion independence: number analyzed (Participants) | 23
  Platelet transfusion independence | 60.9 [38.5 to 80.3]

28. Secondary Outcome: Duration of Post Baseline Transfusion Independence
Description: The duration of transfusion independence is defined as the first time period that a participant received no RBC/platelet transfusions for at least 56 days during the evaluation period.
  Post-baseline transfusion independence is defined as a period of at least 56 days with no RBC or platelet transfusion during the evaluation period. The evaluation period is from the first dose of study drug to the last dose of study drug until the 30 day follow-up visit, disease progression (including clinical progression), or death, whichever was earlier.
Time Frame: as for outcome 26
Population: Enrolled participants who received venetoclax with LDAC at the recommended Phase 2 dose (600 mg) who achieved post-baseline RBC or platelet transfusion independence overall (50), RBC and platelet transfusion independence (37), RBC transfusion independence (39), or platelet transfusion independence (48).
Measure: Median (Full Range); unit: days
Arm/Group | Phase 1+2: 600 mg Venetoclax + LDAC
Number analyzed (Participants) | 50
days
  Duration of RBC and platelet transfusion independence: number analyzed (Participants) | 37
  Duration of RBC and platelet transfusion independence | 150 [56 to 1855]
  Duration of RBC transfusion independence: number analyzed (Participants) | 39
  Duration of RBC transfusion independence | 123 [56 to 1881]
  Duration of platelet transfusion independence: number analyzed (Participants) | 48
  Duration of platelet transfusion independence | 155.5 [56 to 1855]

ADVERSE EVENTS:
Time Frame: All-cause mortality is reported from enrollment through the end of study; maximum time on study was 63.7 months. Adverse events are reported from first dose of study drug until 30 days after last dose of study drug; median (minimum, maximum) duration of treatment was 4.1 (0.2, 62.8) months overall.
Description: All-cause mortality is reported for all enrolled participants. Adverse events are reported for all participants who received at least 1 dose of venetoclax.
Arm/Group | Phase 1: 600 mg Venetoclax + LDAC | Phase 1: 800 mg Venetoclax + LDAC | Phase 2: 600 mg Venetoclax + LDAC
All-Cause Mortality (participants affected / at risk) | 6/8 | 10/10 | 63/76
Serious Adverse Events (participants affected / at risk) | 7/8 | 9/10 | 68/74
Other Adverse Events (participants affected / at risk) | 8/8 | 10/10 | 74/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: 600 mg Venetoclax + LDAC (N=8) | Phase 1: 800 mg Venetoclax + LDAC (N=10) | Phase 2: 600 mg Venetoclax + LDAC (N=74)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (2)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 3 (5) | 22 (34)
HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (2) | 0 (0) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 2 (6)
ATRIOVENTRICULAR BLOCK FIRST DEGREE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
BRADYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
SINUS BRADYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
DIPLOPIA (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
COLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
DIVERTICULUM INTESTINAL HAEMORRHAGIC (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
INTUSSUSCEPTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
LARGE INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
LARGE INTESTINE POLYP (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
ASTHENIA (General disorders) | 1 (1) | 0 (0) | 2 (2)
DEATH (General disorders) | 0 (0) | 0 (0) | 1 (1)
DEVICE RELATED THROMBOSIS (General disorders) | 0 (0) | 0 (0) | 1 (1)
DISEASE PROGRESSION (General disorders) | 0 (0) | 0 (0) | 1 (1)
GAIT DISTURBANCE (General disorders) | 0 (0) | 0 (0) | 1 (1)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 (0) | 0 (0) | 1 (1)
HYPERPYREXIA (General disorders) | 0 (0) | 0 (0) | 1 (1)
MUCOSAL INFLAMMATION (General disorders) | 0 (0) | 0 (0) | 1 (1)
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 0 (0) | 1 (1) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 4 (4) | 2 (2)
SUDDEN DEATH (General disorders) | 0 (0) | 0 (0) | 1 (1)
ACUTE HEPATIC FAILURE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
CHOLECYSTITIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
HEPATIC FAILURE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
BACTERAEMIA (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
BACTERIAL SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
BRONCHOPULMONARY ASPERGILLOSIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
CANDIDA PNEUMONIA (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
CYSTITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
DEVICE RELATED INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 4 (4)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
ESCHERICHIA BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ESCHERICHIA SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 2 (8)
INFECTIOUS PLEURAL EFFUSION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
LARGE INTESTINE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
NOSOCOMIAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OSTEOMYELITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PARAINFLUENZAE VIRUS INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PNEUMOCYSTIS JIROVECII PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 2 (2) | 1 (1) | 11 (14)
PNEUMONIA KLEBSIELLA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PULMONARY SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
RESPIRATORY TRACT INFECTION FUNGAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 8 (10)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
SERRATIA SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 2 (3)
UROSEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
VASCULAR DEVICE INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
INTENTIONAL OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
POST-TRAUMATIC PAIN (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
SKIN LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
SPLENIC RUPTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
SUBDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
AMYLASE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
LIPASE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
TROPONIN INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 1 (1) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
FLUID OVERLOAD (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
BURSITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 5 (5)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
DEMENTIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
HAEMORRHAGIC STROKE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
ISCHAEMIC STROKE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
LACUNAR INFARCTION (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
LETHARGY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
PRESYNCOPE (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
PSYCHOTIC DISORDER DUE TO A GENERAL MEDICAL CONDITION (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
DYSURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
URINARY INCONTINENCE (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (2)
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
PULMONARY ALVEOLAR HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
HYPERTENSION (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: 600 mg Venetoclax + LDAC (N=8) | Phase 1: 800 mg Venetoclax + LDAC (N=10) | Phase 2: 600 mg Venetoclax + LDAC (N=74)
ANAEMIA (Blood and lymphatic system disorders) | 5 (6) | 2 (2) | 19 (72)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 12 (13)
HYPOFIBRINOGENAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 2 (4)
NEUTROPENIA (Blood and lymphatic system disorders) | 4 (10) | 4 (5) | 19 (25)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 4 (4) | 4 (11) | 26 (44)
ANGINA PECTORIS (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 6 (8)
BRADYCARDIA (Cardiac disorders) | 2 (2) | 0 (0) | 2 (3)
CARDIAC FAILURE (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2)
SINUS TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 6 (9)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1) | 6 (6)
HYPERTHYROIDISM (Endocrine disorders) | 1 (1) | 1 (1) | 1 (1)
ERYTHEMA OF EYELID (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
EYE PAIN (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
RETINAL HAEMORRHAGE (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
VISION BLURRED (Eye disorders) | 0 (0) | 0 (0) | 4 (4)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 1 (2) | 11 (17)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (5)
CONSTIPATION (Gastrointestinal disorders) | 2 (3) | 3 (3) | 27 (30)
DIARRHOEA (Gastrointestinal disorders) | 6 (7) | 2 (4) | 34 (61)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 6 (7)
ERUCTATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
FLATULENCE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4)
HAEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
LIP ULCERATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
MOUTH HAEMORRHAGE (Gastrointestinal disorders) | 2 (2) | 0 (0) | 6 (8)
MOUTH ULCERATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (6)
NAUSEA (Gastrointestinal disorders) | 8 (13) | 6 (12) | 48 (67)
ODYNOPHAGIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
PARAESTHESIA ORAL (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 6 (7)
TONGUE HAEMATOMA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (4)
TRICHOGLOSSIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 3 (4) | 3 (5) | 21 (30)
CATHETER SITE INFLAMMATION (General disorders) | 0 (0) | 1 (1) | 0 (0)
CATHETER SITE PAIN (General disorders) | 1 (1) | 1 (1) | 2 (3)
CHEST DISCOMFORT (General disorders) | 1 (1) | 0 (0) | 6 (6)
CHEST PAIN (General disorders) | 1 (2) | 0 (0) | 3 (3)
CHILLS (General disorders) | 1 (1) | 1 (1) | 6 (13)
DEVICE RELATED THROMBOSIS (General disorders) | 1 (1) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 7 (7) | 3 (11) | 28 (52)
INJECTION SITE HAEMATOMA (General disorders) | 1 (1) | 0 (0) | 0 (0)
MALAISE (General disorders) | 1 (1) | 0 (0) | 6 (6)
MUCOSAL INFLAMMATION (General disorders) | 1 (1) | 0 (0) | 8 (9)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1) | 2 (2) | 4 (4)
OEDEMA PERIPHERAL (General disorders) | 2 (5) | 2 (2) | 13 (18)
PAIN (General disorders) | 0 (0) | 0 (0) | 9 (9)
PYREXIA (General disorders) | 1 (3) | 1 (1) | 14 (15)
BRONCHOPULMONARY ASPERGILLOSIS ALLERGIC (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 4 (4)
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 4 (4)
DEVICE RELATED INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 5 (5)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
HERPES SIMPLEX (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
HORDEOLUM (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ORAL CANDIDIASIS (Infections and infestations) | 0 (0) | 1 (1) | 5 (7)
PARONYCHIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 5 (6)
SIALOADENITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 1 (1) | 4 (4)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 7 (9)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 7 (9)
HEAD INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 4 (6)
OVERDOSE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
PERIORBITAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 4 (4)
SUNBURN (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
TOOTH FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
WOUND (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 1 (1) | 0 (0) | 8 (14)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (2) | 1 (5) | 7 (9)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 8 (10)
BLOOD ALBUMIN DECREASED (Investigations) | 0 (0) | 0 (0) | 4 (13)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 (0) | 0 (0) | 10 (27)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 2 (4) | 19 (33)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 1 (7) | 8 (18)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 1 (1) | 0 (0) | 2 (2)
BLOOD URIC ACID INCREASED (Investigations) | 1 (2) | 0 (0) | 1 (1)
HEART RATE IRREGULAR (Investigations) | 1 (1) | 0 (0) | 0 (0)
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 0 (0) | 0 (0) | 8 (11)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 1 (1) | 0 (0) | 0 (0)
LIVER FUNCTION TEST INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
LYMPHOCYTE COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 15 (116)
NEUTROPHIL COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 14 (92)
PLATELET COUNT DECREASED (Investigations) | 1 (1) | 0 (0) | 20 (152)
PROTHROMBIN TIME PROLONGED (Investigations) | 0 (0) | 1 (1) | 1 (1)
SPECIFIC GRAVITY URINE DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
TROPONIN INCREASED (Investigations) | 0 (0) | 0 (0) | 4 (4)
WEIGHT DECREASED (Investigations) | 0 (0) | 0 (0) | 6 (6)
WEIGHT INCREASED (Investigations) | 1 (1) | 1 (1) | 3 (3)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 (0) | 2 (2) | 28 (170)
DECREASED APPETITE (Metabolism and nutrition disorders) | 5 (7) | 2 (2) | 25 (32)
FLUID OVERLOAD (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 3 (4)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (3) | 9 (12)
HYPERMAGNESAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (4)
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 10 (11)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 7 (7)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 10 (28)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 22 (61)
HYPOCHLORAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (4)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 4 (5) | 3 (5) | 36 (77)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1 (2) | 3 (4) | 27 (44)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 16 (48)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 22 (41)
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 12 (20)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 14 (16)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
CHONDROCALCINOSIS PYROPHOSPHATE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 3 (3)
LIMB MASS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (4)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (5)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 4 (4)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 4 (4)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (3) | 11 (13)
CEREBRAL MICROANGIOPATHY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 2 (7) | 1 (1) | 11 (18)
HEADACHE (Nervous system disorders) | 3 (4) | 2 (2) | 20 (24)
LETHARGY (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
PARAESTHESIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
RESTLESS LEGS SYNDROME (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
SINUS HEADACHE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
SOMNOLENCE (Nervous system disorders) | 0 (0) | 0 (0) | 4 (4)
TASTE DISORDER (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
TREMOR (Nervous system disorders) | 0 (0) | 0 (0) | 4 (4)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 11 (11)
CONFUSIONAL STATE (Psychiatric disorders) | 3 (3) | 0 (0) | 7 (7)
DELIRIUM (Psychiatric disorders) | 0 (0) | 0 (0) | 4 (4)
DEPRESSION (Psychiatric disorders) | 1 (2) | 0 (0) | 10 (11)
FLAT AFFECT (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
HALLUCINATION, VISUAL (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
INSOMNIA (Psychiatric disorders) | 1 (1) | 1 (1) | 17 (17)
MOOD ALTERED (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
PROCEDURAL ANXIETY (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
RESTLESSNESS (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0)
SLEEP DISORDER (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 2 (3) | 3 (3) | 6 (10)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 4 (4)
POLLAKIURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 4 (4)
URINARY INCONTINENCE (Renal and urinary disorders) | 0 (0) | 0 (0) | 4 (4)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 19 (24)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 20 (33)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (3)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 9 (12)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 7 (7)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 4 (4)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 9 (10)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (2) | 10 (10)
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 4 (4)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
ACNE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 6 (6)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
NAIL DISCOLOURATION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
PETECHIAE (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 7 (14)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 10 (11)
PURPURA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 7 (8)
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2)
RASH MACULAR (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 5 (5)
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
SKIN LESION (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2)
STASIS DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
HAEMATOMA (Vascular disorders) | 1 (1) | 1 (1) | 2 (2)
HYPERTENSION (Vascular disorders) | 1 (3) | 1 (1) | 14 (19)
HYPOTENSION (Vascular disorders) | 2 (2) | 2 (3) | 12 (14)
MACROANGIOPATHY (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-10-22): https://cdn.clinicaltrials.gov/large-docs/33/NCT02287233/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-02): https://cdn.clinicaltrials.gov/large-docs/33/NCT02287233/SAP_001.pdf